CLINICAL TRIAL: NCT03636646
Title: Analysis of the Posterior Wall Fracture of the Acetabulum
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hamada Mohamed Kamel, Dr, Assiut University
Other Study IDs: Posterior wall fracture
Record Dates: First submitted 2018-08-15; First posted 2018-08-17 (Actual); Last update posted 2018-08-17 (Actual); Status verified 2018-08

CONDITIONS: Acetabular Fracture

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: X.ray — Surgical treatement of posterior acetabular wall fractures

SUMMARY:
Assessement,evaluation of postoperativ reduction of posterior wall acetabular fractures in Assiut University Hospital

DETAILED DESCRIPTION:
Posterior wall fracture of the acetabulum resemble 30% of acetabular fracture,surgical treatement is the 1st choice now for most of these fractures as it aimes to restore joint conjuroity and decreases the possibelities of osteoarthrities of the hip joint,in this study investigators will make analysis and assessement of the quality of postoperative reduction which is the main indicator of outcome of acetabular fractures in adult patients in Assiut University Hospitsls

ELIGIBILITY:
Inclusion Criteria:

* adult patients of both sexes with posterior acetabular wall fracture either isolated or associated with other fractures

Exclusion Criteria:

* other types of acetabular fractures not associated with posterior wall fracture

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients of both sexes with posteriir acetabular wall fractures
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2018-08 (Estimated); Primary Completion 2019-04 (Estimated); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
Analysis of the posterior wall fractures of the acetabulum | Basline
  Analysis and assessement of the quality of postoperative reduction of posterior wall fractures of the acetabulum using postoperative x.ray by MATTA Score

IPD SHARING:
Plan to Share IPD: Undecided